CLINICAL TRIAL: NCT04367350
Title: Prospective Registry for Multimodal Assessment of Neuromuscular Pathology Associated With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Brief Title: Prospective Registry of Corona Virus Disease 2019 (Covid-19) Patients With Neuromuscular Involvement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 246/2020BO2
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COVID; Sars-CoV2; Corona Virus Infection; Myositis; Myocarditis
MeSH Terms: conditions — Coronavirus Infections; Myositis; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laboratory biomarkers — creatine kinase, troponin, urine myoglobin, and autoimmune antibodies
Diagnostic Test: muscle ultrasound — Muscle echogenicity in the upper and lower extremities, the accessory respiratory serratus anterior muscle, and abdominal wall according to qualitative ultrasound assessment (Heckmatt score)

SUMMARY:
Prospective registry for multimodal assessment of neuromuscular pathology associated with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, enrolling consecutive patients with corona virus disease 2019 (Covid-19), who are admitted to the intensive care unit of the department of anesthesiology and intensive care medicine, or the department of neurology at Tübingen University Hospital.

DETAILED DESCRIPTION:
The prospective registry shall provide new insights into muscular involvement associated with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. For that reason consecutive patients with proven corona virus disease 2019 (Covid-19), who are admitted to the intensive care unit of the department of anesthesiology and intensive care medicine, or the department of neurology at Tübingen University Hospital, are enrolled. Multimodal assessment of neuromuscular pathology is based on medical history, laboratory biomarkers including inflammation parameters and autoimmune antibodies, vital parameters monitoring, muscle ultrasound, transthoracic echocardiography, electroneurography, as well as electromyography. Inclusion of follow-up visits permit longitudinal and prognostic evaluation of diagnostic and therapeutic interventions (e.g. immunomodulation with immunoglobulins, corticosteroids, or interleukin 6 receptor antagonists).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Proven severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection

Exclusion Criteria:

* active or known history of myopathy or advanced stage neuropathy
* refusal to participate in clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with corona virus disease 2019 (Covid-19), who are admitted to the intensive care unit of the department of anesthesiology and intensive care medicine, or the department of neurology at Tübingen University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of elevated creatine kinase in hyperacute phase | 1 week
  Elevation of creatine kinase during hyperacute phase of corona virus disease 2019 (Covid-19)

SECONDARY OUTCOMES:
Rate of elevated creatine kinase | 24 months
  Elevation of creatine kinase during hyperacute, acute, subacute and chronic phase of corona virus disease 2019 (Covid-19)
Rate of two-peak elevation of creatine kinase during acute phase | 30 days
  Two-peak elevation of creatine kinase during acute phase of corona virus disease 2019 (Covid-19)
Rate of myositis-specific antibodies | 24 months
  Presence of myositis-specific antibodies on admission, at two weeks, and at end of follow-up
Rate of antimyocardial antibodies | 24 months
  Presence of antimyocardial antibodies on admission, at two weeks, and at end of follow-up
Area under the curve (AUC) of elevated creatine kinase | 24 months
  Level of creatine kinase elevation in the hyperacute, acute, subacute and chronic phase of corona virus disease 2019 (Covid-19) assessed by the area under the curve (AUC)
Peak-levels of elevated creatine kinase | 24 months
  Maximal value of creatine kinase elevation in the hyperacute, acute, subacute and chronic phase of corona virus disease 2019 (Covid-19)
Peak-levels of troponin | 30 days
  Maximal value of troponin in the acute phase of corona virus disease 2019 (Covid-19)
Peak-levels of urine myoglobin | 30 days
  Maximal value of urine myoglobin in the acute of corona virus disease 2019 (Covid-19)
Rate of muscle hyperechogenicity | 24 months
  Muscle hyperechogenicity in the upper and lower extremities, the accessory respiratory serratus anterior muscle, and abdominal wall according to qualitative ultrasound assessment (Heckmatt score) during the hyperacute, acute, subacute and chronic phase of corona virus disease 2019 (Covid-19)
Peak-muscle hyperechogenicity | 24 months
  Peak-muscle hyperechogenicity in the upper and lower extremities, the accessory respiratory serratus anterior muscle, and abdominal wall according to qualitative ultrasound assessment (Heckmatt score) during the hyperacute, acute, subacute and chronic phase of corona virus disease 2019 (Covid-19)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided